CLINICAL TRIAL: NCT00001018
Title: Blinded, Placebo-Controlled, Single-Dose Pharmacokinetics and Dose Escalation, Efficacy, and Safety Study of Letrazuril for AIDS-Related Cryptosporidial Diarrhea
Brief Title: A Study of Letrazuril in the Treatment of AIDS-Related Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Janssen Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: ACTG 198; Protocol JRD 65731/1001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-10

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Cryptosporidiosis; Diarrhea; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; Triazines
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — letrazuril

INTERVENTIONS:
Drug: Letrazuril

SUMMARY:
To determine the pharmacokinetic profile of single doses of letrazuril in patients with AIDS-related cryptosporidial diarrhea; to determine the dose proportionality of single escalating doses of letrazuril; to determine steady-state concentrations of letrazuril; to evaluate the safety and efficacy of escalating doses of letrazuril, compared with placebo, for patients with AIDS-related cryptosporidial diarrhea.

Letrazuril, the p-fluor analog of diclazuril, has been shown in an animal model to prevent infections by organisms closely related to the intracellular parasite Cryptosporidium. Reliable data are needed to show the effectiveness of letrazuril in treating AIDS-related cryptosporidial diarrhea.

DETAILED DESCRIPTION:
Letrazuril, the p-fluor analog of diclazuril, has been shown in an animal model to prevent infections by organisms closely related to the intracellular parasite Cryptosporidium. Reliable data are needed to show the effectiveness of letrazuril in treating AIDS-related cryptosporidial diarrhea.

Four groups of eight patients receive escalating doses of oral letrazuril (or placebo). In each group, six patients are randomized to receive letrazuril and two patients receive matching placebo. In the pharmacokinetics determination phase of the study, patients receive a single dose of letrazuril or placebo following a meal. Following a 72-hour blood collection, patients enter the blinded, treatment phase of the study and receive letrazuril or placebo as a single dose daily, after a meal, for 3 weeks. Patients with persistent Cryptosporidium oocysts in their stools at the end of the blinded treatment phase may continue with open-label treatment of letrazuril at the same dose for 4 weeks; the dose may subsequently be escalated every 4 weeks, to a maximum, if oocysts persist. Patients who have Cryptosporidium oocysts eradicated from their stools will discontinue treatment and be followed for 3 months. All patients undergo clinical follow-up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Anti-diarrheal and antiemetic medications.
* Anti-HIV agents such as zidovudine, ddI, and ddC if dosing regimens were stable for at least 3 weeks prior to start of study drug.

Patients must have:

* AIDS.
* Chronic diarrhea with presence of Cryptosporidium oocysts in a stool specimen.
* CD4 count < 150/mm3 (not required if patient has had cryptosporidiosis for a minimum of 4 weeks).
* Life expectancy of at least 1 month.

Prior Medication:

Allowed:

* Anti-HIV agents such as zidovudine, ddI, and ddC if dosing regimens were stable for at least 3 weeks prior to start of study drug.
* Anti-diarrheal and antiemetic medications.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Grade 4 hematologic toxicity or grade 3 other toxicity ( patients with grade 3 hepatic toxicity may be enrolled if abnormalities are considered to be caused by biliary cryptosporidiosis).
* Presence of other diarrhea-causing pathogens.
* Active (defined as newly diagnosed, progressive, or requiring therapeutic intervention) opportunistic infection that requires antimicrobial therapy (patients receiving maintenance or prophylactic antimicrobial therapy for opportunistic infection may be enrolled if the dosing regimen has been stable for at least 3 weeks).
* Evidence of cytomegalovirus retinitis or colitis.

Concurrent Medication:

Excluded:

* Ganciclovir, cancer chemotherapy, or interferon-alpha or other immunomodulating agents.
* Any investigational drug (drugs available under an FDA-authorized expanded access program will not be considered investigational).

Prior Medication:

Excluded:

* Any investigational drug within 1 month prior to start of study drug (drugs available under an FDA-authorized expanded access program will not be considered investigational).
* Ganciclovir, cancer chemotherapy, or interferon-alpha or other immunomodulating agents within 7 days prior to start of study drug.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Overall Officials: Moskovitz BL, Study Chair
Locations (4):
- United States (4):
  - USC School of Medicine, Los Angeles, California
  - Dr Douglas Dieterich, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York

REFERENCES:
- [Background] Guillem S, Gomez M, Romeu J, Raventos A, Fernandez A, Condom MJ, Clotet B. Letrazuril for the treatment of severe cryptosporidial diarrhoea in AIDS. Int Conf AIDS. 1992 Jul 19-24;8(2):B129 (abstract no PoB 3257)
- [Background] Harris M, Deutsch G, MacLean JD, Tsoukas CM. A phase I study of letrazuril in AIDS-related cryptosporidiosis. AIDS. 1994 Aug;8(8):1109-13. doi: 10.1097/00002030-199408000-00011. PMID 7986407
- [Background] Rubbert A, Schwab J, Kalden JR, Nusslein H. Myositis, fever, rash and thrombopenia after letrazuril treatment of intestinal cryptosporidiosis: a case report. Int Conf AIDS. 1993 Jun 6-11;9(1):373 (abstract no PO-B10-1430)